CLINICAL TRIAL: NCT05082103
Title: Effect of Enzyme-containing Lozenges on Dental Biofilm Accumulation in Healthy Individuals: A Randomized Placebo-controlled Clinical Trial
Brief Title: Effect of Enzymes on Dental Biofilm Accumulation in Healthy Individuals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated after interim data analysis
Sponsor: Novozymes A/S (Industry)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NZ-OHBFC-2021-01
Record Dates: First submitted 2021-09-16; First posted 2021-10-18 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Dental Plaque
Keywords: Enzymes; Dental plaque; Gingivitis; Oral microbiome
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enzyme lozenge 1 (Active Comparator): The lozenge contains three plaque extracellular matrix degrading enzymes
  Interventions: Other: Enzyme lozenge 1
- Enzyme lozenge 2 (Active Comparator): The concentration of the three enzymes in the "Enzyme lozenge 2" is threefold the enzyme concentration than in the "Enzyme lozenge 1"
  Interventions: Other: Enzyme lozenge 2
- Placebo lozenge (Placebo Comparator): The placebo lozenge contains the same ingredients except for the enzymes and has an identical taste, color and texture
  Interventions: Other: Placebo lozenge

INTERVENTIONS:
Other: Enzyme lozenge 1 — Participants are instructed to take one enzyme containing lozenge three times daily, at least 30 min after a meal, for 14 days. No normal oral hygiene procedures are allowed during the intervention period.
  Arms: Enzyme lozenge 1
Other: Enzyme lozenge 2 — Participants are instructed to take one lozenge with 3x higher enzyme concentration three times daily, at least 30 min after a meal, for 14 days. No normal oral hygiene procedures are allowed during the intervention period.
  Arms: Enzyme lozenge 2
Other: Placebo lozenge — Participants are instructed to take one placebo lozenge three times daily, at least 30 min after a meal, for 14 days. No normal oral hygiene procedures are allowed during the intervention period.
  Arms: Placebo lozenge

SUMMARY:
The purpose of the study is to assess the effect of enzyme containing lozenges on dental plaque accumulation in healthy adults.

DETAILED DESCRIPTION:
The purpose of the study is to examine the clinical effects of lozenges containing three extracellular matrix-degrading enzymes on dental plaque accumulation and removal, prevention of gingivitis, and oral microbiome composition after professional tooth cleaning, as compared to a placebo lozenge without enzymes. Two different concentrations of the enzymes will be tested, to investigate a potential dose-dependent effect of the enzymes. Furthermore, safety of the enzyme lozenge will be assessed by clinical evaluation of the oral mucosa. The null hypothesis is that treatment with enzyme-containing lozenges does not affect plaque accumulation as compared to a placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy males and females ≥18 years of age.
* Able to read, sign and receive a copy of the signed informed consent form.
* Have at least 20 natural teeth.

Exclusion Criteria:

* Clinically visible active caries lesions and/or periodontitis.
* Significant oral soft tissue pathology based on a visual examination.
* History of allergy or significant adverse events following use of oral hygiene products such as toothpastes, mouth rinses, breath mints, lozenges, or chewing gum or their ingredients.
* History of allergies to ingredients in the test product.
* Self-reported as pregnant or nursing.
* Self-reported serious medical conditions.
* Antibiotic or anti-inflammatory medication within 30 days of screening visit.
* Orthodontic appliances, including retainers, peri/oral piercings, or removable partial dentures.
* Acute sinusitis or severe oral-pharyngeal infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Plaque amount | Change in QHPI score from baseline to 24 hours' follow-up
  Dental plaque accumulation after 1-day use of either a test or placebo investigational lozenge assessed by the Turesky modified Quingly-Hein Plaque Index (QHPI) (score 0-5, 0 being no plaque, 5 being entire tooth covered with plaque)

SECONDARY OUTCOMES:
Plaque amount | Change in QHPI score from baseline to Day 7 follow-up and from baseline to Day 14 follow-up
  Dental plaque accumulation after 7 and 14 days assessed by the Turesky modified Quingly-Hein Plaque Index (QHPI) (score 0-5, 0 being no plaque, 5 being entire tooth covered with plaque)
Gingivitis | Change in GI from baseline to Day 14 follow-up
  Development of gingivitis after 14 days assessed by the Gingival Index of Löe and Silness (GI) (score 0-3, 0 being no gingivitis, 3 being excessive gingivitis)
Plaque removal | Day 14 visit
  Plaque removal by mechanical treatment with a water-/airpik. The technique will be applied professionally at the clinical site by co-investigator.
Oral microbiome | Change in microbiome composition from baseline to Day 14 follow-up
  Oral microbiome composition
Plaque fluorescence intensity measurement | Change in intensity measurement from baseline to Day 7 follow-up and Day 14 follow-up
  Dental plaque accumulation assessed by fluorescence intensity measurements, to provide information on the individual level of plaque formation. Soft biofilm on the teeth is calculated using an appropriate software program, compatible with the device used.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Rose Jørgensen, DDS, PhD, Study Director — Novozymes A/S; Sebastian Schlafer, DDS, PhD, Principal Investigator — Aarhus University, Department of Dentistry and Oral Health
Locations (1):
- Aarhus University, Department of Dentistry and Oral Health, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rikvold PD, Johnsen KK, Del Rey YC, Hansen LBS, Knap I, Holz C, Meyer RL, Jorgensen MR, Schlafer S. The Effect of Enzymes on Dental Plaque: A Randomized Controlled Trial. J Dent Res. 2026 Feb;105(2):236-244. doi: 10.1177/00220345251347959. Epub 2025 Jul 17. PMID 40676928